CLINICAL TRIAL: NCT03003715
Title: Brain as a Therapeutic and Research Target in Trigeminal Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alexandre DaSilva, DDS, MS, DDS, D.Med.Sc., University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00024607
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Trigeminal Neuropathic Pain
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Refractory Trigeminal Neurpathic Pain (TNP) Patients (Experimental): All patients receive QST prior to PET scan used to obtain baseline measures, then placebo tDCS, followed by QST and Active tDCS, over the course of a 90 minute PET scan; QST is used again to take final measurements 30 minutes later.
  Interventions: Procedure: PET Scans; Procedure: transcranial direct current stimulation (tDCS); Procedure: MRI; Other: sham tDCS (prior to real tDCS)
- Healthy volunteers (Experimental): All volunteers receive QST prior to PET scan used to obtain baseline measures, then placebo tDCS, followed by QST and Active tDCS, over the course of a 90 minute PET scan; QST is used again to take final measurements 30 minutes later.
  Interventions: Procedure: PET Scans; Procedure: transcranial direct current stimulation (tDCS); Procedure: MRI; Other: sham tDCS (prior to real tDCS)

INTERVENTIONS:
Procedure: PET Scans — Two 90 minute scans whose maximum radiological dose is 15 mCi [11 C] carfentanil, a selective and specific mu-opioid receptor radioligand. The first one provided baseline data, and the second occurred with the sequence of sham tDCS and tDCS as described in each arm description.
Procedure: transcranial direct current stimulation (tDCS) — In active tDCS, a 2 milli-amp transcranial direct current stimulation is for 20 minutes.
Procedure: MRI — No radiotracer is used; 3 tesla scanner; all participants have MRI prior to PET scans.
Other: sham tDCS (prior to real tDCS) — For sham tDCS, current is applied only for 30 seconds, as sensations arising from tDCS treatment occur only at the beginning of application; however the equipment will be on the participant for 20 minutes to match that of the active tDCS application.

SUMMARY:
The main goal of this study to integrate techniques producing images of the brain (also called neuroimaging techniques) with non-invasive brain stimulation to investigate factors that may be associated with chronic pain in patients with Trigeminal Neuropathic Pain (TNP).

DETAILED DESCRIPTION:
Trigeminal neuropathic pain (TNP) disorders, such as classical trigeminal and post-surgical neuralgia, are debilitating chronic conditions with pain that is either spontaneous or that can be intensely evoked by light touch to the facial skin. Although neuroimaging techniques have provided insights into some brain mechanisms of experimental trigeminal pain in humans (DaSilva et al., 2002; Borsook et al., 2003), it is not well understood how structural and molecular mechanisms are affected during the course of TNP, and how they can be safely modulated for therapeutic and research purposes. Understanding these processes is crucial to determine the structures engaged in the development and persistence of TNP.

We will test the hypothesis that chronicity of TNP is sustained by changes at cellular and molecular levels in neural circuits associated with pain perception and modulation, rather than by the initial peripheral etiology, and that this dysfunction can be safely targeted and modulated as a therapeutic approach by transcranial direct current stimulation (tDCS). To achieve this goal we will use a neuroimaging technique, PET, employing a mathematical model that permits the quantification of opioid receptor availability in vivo.

ELIGIBILITY:
Patient Inclusion Criteria:

* Daily chronic TNP for at least 6 months not adequately controlled by pervious medicine therapies;
* minimal average baseline pain score of 4 (moderate to severe) in the visual analogue scale (VAS);
* unilateral pain
* orofacial allodynic region to mechanical (light touch or palpation) or thermal stimulation (head or cold);

Patient Exclusion Criteria:

* pregnancy or planning to become pregnant
* local pathology (e.g. orofacial lesion)
* history of systemic disorders (e.g. MS)
* history of other chronic pain disorder (e.g. back pain)
* recent orofacial surgery or trauma (< 6 months)
* history of central origin disorders (e.g. stroke)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in MOR BPND levels | place weeks after not more than 6months
  change from baseline to versus sham or active tDCS

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre F DaSilva, DMedSci, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States